CLINICAL TRIAL: NCT03763110
Title: Evaluation of Post-Operative Pain After Regenerative Endodontic Using Photo-Activated Oral Disinfection Versus Triple-Antibiotic Paste for Management of Necrotic Young Permanent Anterior Teeth
Brief Title: Photo-Activated Disinfection Versus Triple-Antibiotic Paste for Management of Necrotic Young Permanent Anterior Teeth
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, ElShaimaa Abdelhafiz Abdelrahim, assistant lecturer in paediatric dentistry department at Fayoum university, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Regenerative endodontic
Record Dates: First submitted 2018-11-17; First posted 2018-12-04 (Actual); Last update posted 2018-12-05 (Actual); Status verified 2018-08

CONDITIONS: Pulp Necrosis
MeSH Terms: conditions — Dental Pulp Necrosis | interventions — Photochemotherapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Photo Activated Disinfection (Experimental): Photoactivated disinfection (PAD) is based on the interaction of a photosensitive antibacterial agent and a light source. It uses a nontoxic dye [named photosensitizer PS] and low-intensity visible light. In oxygen presentation, these combine to produce some cytotoxic species. The PS molecules attach to bacteria membrane
  Interventions: Device: Photo Activated Disinfection
- Antibiotic paste (Active Comparator): Hoshino et al. recommended a ratio of 1:1:1 of metronidazole (500 mg), minocycline (100 mg) and ciprofloxacin (200 mg) for the 3Mix formulation
  Interventions: Drug: antibiotic paste

INTERVENTIONS:
Device: Photo Activated Disinfection — Photoactivated disinfection (PAD) is based on the interaction of a photosensitive antibacterial agent and a light source. It uses a nontoxic dye [named photosensitizer PS] and low-intensity visible light. In oxygen presentation, these combine to produce some cytotoxic species. The PS molecules attach to bacteria membrane
  Other Names: Photodynamic therapy (PDT)
  Arms: Photo Activated Disinfection
Drug: antibiotic paste — An antibiotic mixture composed of ciproﬂoxacin, metronidazole, and minocycline, known as triple antibiotic paste (TAP) or "3mix", has been the most widely used medicament, This goes back to the studies by Hoshino et al.1996
  Other Names: Triple antibiotic paste
  Arms: Antibiotic paste

SUMMARY:
This study aims to compare regenerative endodontics for necrotic young permanent anterior teeth using oral photo-activated disinfection versus triple antibiotic paste in terms of:

1. Clinical success in terms of absence of any complication such as spontaneous pain, sinus or swelling.
2. Radiographic success in terms of healing of periapical radiolucency or increase root thickness, length or apical closure.

DETAILED DESCRIPTION:
Disinfection of the root canal system is thought to be critical to the success of Regenerative Endodontic Procedures (REPs) as infection prevents regeneration, repair and stem cell activity . A suitable material for using as intra-canal medicament seems to be antibiotic. Triple antibiotic paste (TAP) containing metronidazole, ciprofloxacin and minocycline has been reported to be a successful regimen in controlling the root canal pathogen and in managing necrotic young permanent tooth .

Recently, new disinfection methods have been developed to overcome the limitations of conventional disinfecting protocols that they may neither reduce the number of bacteria to a satisfactory level nor minimize the toxicity to periapical stem/progenitors . Other concerns regarding the use of TAP are tooth discoloration after treatment and bacterial resistance. Photo-activated oral disinfection is a novel disinfection method which present a great solution for the problem associated with triple antibiotic paste

ELIGIBILITY:
Inclusion Criteria:

* Healthy children with no physical, mental or systemic conditions.
* Developmental age of the child is the most important factor so periapical x- ray will be taken first to assure apex immaturity.
* No sex predilection.
* Restorable necrotic young permanent anterior teeth

Exclusion Criteria:

* Root fracture.
* Internal or external root resorption.
* Parents or guardians refuse to participate in the study.

Ages: 8 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2016-10-15 (Actual); Primary Completion 2018-12-15 (Estimated); Study Completion 2019-04-15 (Estimated)

PRIMARY OUTCOMES:
absence of postoperative pain | immediate post operative
  binary question by asking patients (yes or no)
absence of postoperative pain | at 3 months follow up
  binary question by asking patients (yes or no)
absence of postoperative pain | at 6 months follow up
  binary question by asking patients (yes or no)
absence of postoperative pain | at 9 months follow up
  binary question by asking patients (yes or no)
absence of postoperative pain | at 12 months follow up
  binary question by asking patients (yes or no)

SECONDARY OUTCOMES:
healing of sinus | immediate post operative, 3 months, 6 months, 9 months, 12 months
  Clinical success in term of absence of sinus (Yes or No)
healing of swelling | immediate post operative, 3 months, 6 months, 9 months, 12 months
  Clinical success in term of absence of swelling (Yes or No)
healing of periapical radiolucency | baseline, 6 months, 12 months
  Radiographic success in term of healing of periapical or radiolucency (Yes or No)
change in root length | baseline, 6 months, 12 months
  Radiographic evaluation by calibration of root length in millimetre by Digora
change in dentin root thickness | baseline, 6 months, 12 months
  Radiographic evaluation by calibration of root thickness in millimetre by Digora
change in apical diameter | baseline, 6 months, 12 months
  Radiographic evaluation by calibration of apical diameter in millimetre by Digora